CLINICAL TRIAL: NCT04864431
Title: The Effect of Vitamin D on Factors Contributing Pre Cachexia and Cachexia, a Study on Epithelial Ovarian Cancer
Brief Title: Vitamin D and Pre Cachexia and Cancer Cachexia in Epithelial Ovarian Cancer
Acronym: VitD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Collaborators: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Principal Investigator, dr. Nurul Ratna Mutu Manikam, M.Gizi., Sp.GK, Principle Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VitDCaOV
Record Dates: First submitted 2021-04-11; First posted 2021-04-28 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Vitamin D; Pre cachexia; Cachexia; Epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Cachexia | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Intervention group: vitamin D 2000 IU ; Control group: placebo
Who Masked: Participant, Investigator
Masking Description: Neither do investigator nor participants will not know the random allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Active Comparator): Daily vitamin D3 2000 IU on day 1 through day 180 Intervention: vitamin D3 2000 IU
  Interventions: Dietary Supplement: Vitamin D
- Control group (Placebo Comparator): Daily placebo (saccharum lactis) on day 1 through day 180 Intervention: placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D capsules: each capsule contain 2 tablets of vitamin D 1000 IU. One capsule will be taken on day 1 through 180
  Other Names: cholecalciferol
  Arms: Vitamin D group
Other: Placebo — Placebo capsule: Each capsule contain saccharum lactis. One capsule will be taken on day 1 through 180
  Arms: Control group

SUMMARY:
Several ex vivo, in vitro, and observational studies on various type of cancer shown positive effect of vitamin D. Vitamin D has widely known as immunomodulator property in various diseases. However, it remains limited studies on immunity and cachexia in cancer, particularly in ovarian cancer. This study will investigate the effect of vitamin D in immune response during chemotherapy among epithelial ovarian cancer patients who have a low level of vitamin D and cachexia

DETAILED DESCRIPTION:
Studies result from laboratory suggested that vitamin D inhibit cancer cell proliferation and upregulate apoptosis pathway. Data from observational and ecology studies showed the inverse relationship between level of vitamin D and cancer risk. Clinical trials on colorectal, prostate, and breast cancer suggested that vitamin D had positive effect and improved clinical markers.

Vitamin D may alter immune response through regulation on cytotoxic CD8 T-lymphocyte and reduce pro inflammatory cytokines. High level of interleukin-6 and other cytokines in cancer may decrease lymphocyte T activity, resulting lowering effect of immune response.

This clinical trial will enroll 54 adults with newly diagnosed epithelial ovarian cancer patients. Following receive of informed consent, they will randomly allocated to receive whether vitamin D 2000 IU or placebo during chemotherapy period (6 cycles).

Subjects will fill out questionnaire on their first visit as well as each chemotherapy cycle (each month). Questionnaire will ask about demographic data, meal intake, sun exposure, and cachexia questionnaire (based on Cachexia Score). Subjects will also be examined on their physical status, anthropometry (weight, height, waist circumference), as well as body composition (fat mass, fat free mass, fat free mass index, phase angle).

Blood samples will be drawn from peripheral vein and sent to National Cancer Referral Hospital laboratory to measure 25(OH)D level, interleukin-6, CD8 cytotoxic level, CD8 cytotoxic activity, and circulating tumor cells. Blood collection will be done on the first visit, 3rd cycle of chemotherapy, and last cycle of chemotherapy. Subjects will be given their samples result during follow-up visit.

Vitamin D3 (Prove D3®) is donated from PT. Kalbe Farma. Departement of Medicine Physic Indonesia University as the third party which provides randomization and capsules containing vitamin D and placebo. Randomization key will be opened by the third party after finishing statistical data analysis. This study is being submitted a grant from Kalbe-BRIN.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-60 years old who are newly diagnosed with ovarian cancer based on histopathology
2. epithelial ovarian cancer stage II-III
3. haven't received chemotherapy
4. pre-cachexia or cachexia
5. level of vitamin D below 30 ng/ml
6. no vitamin D allergy
7. ability and willingness to understand and provide informed consent

Exclusion Criteria:

1. autoimmune disease
2. chronic liver disease
3. chronic renal disease
4. known had hypercalcemia
5. refractory cachexia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of immune response in participants receiving vitamin D change from baseline as assessed by lymphocyte CD8 | 6 months
  lymphocyte CD8 is measured by flowcytometry

SECONDARY OUTCOMES:
Find the change of vitamin D level | 6 month
  vitamin D level is measured by Electro-Chemiluminescence Immunoassay (e CLIA). The normal range is 30-100 ng/ml
Find the daily intake of vitamin D from food | 1 month
  The amount of vitamin D intake from food in one month is analyzed using food frequency questionnaire in microgram unit measurement. To find the daily intake from food is calculated the total intake in 1 month divided by 30 days. Recommended daily allowance of vitamin D intake from food is 15 microgram/day
Find the rate of sun exposure | 1 week
  sun exposure defined as total duration of sun exposure per day. It assessed using "sun exposure questionnaire". It is calculated based on time outdoor multiply by amount of skin exposure (face, hand, arm, leg, sun bathing), added up everyday for one week. The minimum score is 0 and the maximum score is 56. No score is defined as either adequate or inadequate exposure
Effect of vitamin D in lowering inflammation | 6 months
  defined inflammation as interleukin-6 which is measured by enzyme-linked immunosorbent assay in ng/ml unit measurement. Interleukin-6 increases if the level more than 4 pg/ml
Effect of vitamin D in lowering circulation tumor cells (CTC) | 6 months
  the number of tumor cells in blood. Positive CTC if there are 5 tumor cells in 7,5 ml of blood
Effect of vitamin D in improving staging of cachexia | 6 month
  a diagnostic tools for staging cachexia is measured by Cachexia Score (CASCO). The components of CASCO are body weight loss and composition, inflammation/metabolic disturbances, physical performance, anorexia, and quality of life. CASCO score is presented by numerical scale and classified as mild (score 0-25), moderate (26-50), severe (51-75), and terminal (76-100)

CONTACTS AND LOCATIONS:
Overall Officials: Nurul Ratna Mutu Manikam, MD, MSc, Principal Investigator — Indonesia University
Locations (3):
- Indonesia (3):
  - Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta
  - Tarakan Hospital, Jakarta Pusat, Jakarta Special Capital Region
  - Dharmais National Cancer Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No
Details will be provided at a later date